CLINICAL TRIAL: NCT01699399
Title: A Randomized, Controlled Trial Comparing Water Exchange, Water Immersion and Air Insufflation Methods During Colonoscopy With the Option of on Demand Sedation
Brief Title: Comparing Water Exchange, Water Immersion and Air Insufflation Methods During Colonoscopy With the Option of on Demand Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Chief of department of gastroenterology and hepatology, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DTCRD101(2)-E-03
Record Dates: First submitted 2012-09-30; First posted 2012-10-03 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Colon Neoplasm
Keywords: colonoscopy; pain; sedation; water
MeSH Terms: conditions — Colonic Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- water immersion (Experimental): infuse water during insertion phase of colonoscopy instead of air insufflation; remove the water during withdrawal phase.
  Interventions: Procedure: water immersion
- water exchange (Experimental): infuse and remove water during the insertion phase of colonoscopy. Air insufflation is used only in the withdrawal phase
  Interventions: Procedure: water exchange
- air insufflation (Active Comparator): standard colonoscopy using traditional air insufflation during insertion
  Interventions: Procedure: air insufflation

INTERVENTIONS:
Procedure: water immersion
  Arms: water immersion
Procedure: water exchange
  Arms: water exchange
Procedure: air insufflation
  Arms: air insufflation

SUMMARY:
This prospective, randomized controlled trial compares traditional air insufflation with water immersion and water exchange in patients undergoing colonoscopy using on demand sedation. We test the hypothesis that compared with air insufflation the proportion of patients who require on demand sedation during colonoscopy will be significantly lowered by water immersion and water exchange, and water exchange will produce the greatest reduction

DETAILED DESCRIPTION:
The patients will be allocated into 3 groups by computerized randomization. In group A (water exchange), water will be infused and removed at the same time throughout the entire colon during the insertion phase with the air pump turned off. In group B (water immersion), water will be infused in the insertion phase and removed in the withdrawal phase. The water will be used mainly to open the lumen, without attempting to clear the colon contents. In group A and B, warm-to-touch water will be infused mainly infused through the accessory channel of the colonoscope using a foot-switch controlled water pump (JW2, Fujinon, Saitama, Japan). Air insufflation not used until the cecum has been reached. . In group C, air insufflation will be used throughout the procedure. Aliquots of 30 to 50 ml of water will be used for washing residual stool, as needed. In all three groups, loop reduction maneuvers, abdominal compression and change of patient position will be utilized at the discretion of the colonoscopist and recorded. Intubation of the cecum will be defined as successful only if the base of the cecum is touched with the tip of the colonoscope. Detailed examinations will be undertaken during the withdrawal phase.

During colonoscopy, a study nurse will ask the patient to report the level of pain (0 = none, 10 = most severe) at 2 to 3-minute intervals or at any time the patient voiced discomfort. For pain scores ≧2, maneuvers to minimize pain will be implemented. Immediately thereafter, the nurse will offer sedation, which the patients can accept or decline. If accepted, after an initial bolus of 1 mg/kg or 0.5 mg/kg for patients over 65 years propofol (Diprivan, Astra-Zeneca, Stockholm, Sweden) will be titrated in 20- to 30-mg increments to achieve an adequate level of sedation. The need of additional drug will be estimated by patient pain response (moans, grimaces and movements). Usually no more propofol will be added during the withdrawal phase. The initial amount of propofol, and those before and after arrival to the cecum will be recorded.

The following parameters will be evaluated and recorded on the patient data sheet: quality of bowel preparation, cecal intubation time, withdrawal time total procedure time, use of abdominal pressure, need for changing position, presence of polyps and reasons for incomplete colonoscopy.

The procedure will be recorded and stored as digital files.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy performed by the endoscopist at our endoscopic suite

Exclusion Criteria:

* request for sedation, indicated for bidirectional endoscopy, obstructive lesions of the colon, allergy to meperidine or propofol, American Society of Anesthesiology (ASA) risk Class 3 or higher, massive ascites, past history of partial colectomy, or refusal to provide written informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Proportions of patients requiring sedation | 3 months

SECONDARY OUTCOMES:
patient pain during insertion | 3 months

OTHER OUTCOMES:
post-procedure discomforts and 30 days complication rate | one month
  telephone follow up for post-procedure discomforts and 30 days complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, M.D., Principal Investigator — Dalin Tzu Chi General Hospital
Locations (1):
- Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Hsieh YH, Lin HJ, Tseng KC. Limited water infusion decreases pain during minimally sedated colonoscopy. World J Gastroenterol. 2011 May 7;17(17):2236-40. doi: 10.3748/wjg.v17.i17.2236. PMID 21633535
- [Background] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405
- [Background] Radaelli F, Paggi S, Amato A, Terruzzi V. Warm water infusion versus air insufflation for unsedated colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2010 Oct;72(4):701-9. doi: 10.1016/j.gie.2010.06.025. PMID 20883846